CLINICAL TRIAL: NCT05623969
Title: Markers of Atrial Cardiopathay
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Zarief Farhan, principal investigator, Assiut University
Other Study IDs: atrial cardiopathay
Record Dates: First submitted 2022-11-02; First posted 2022-11-21 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Atrial Cardiopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Holter ,Echo , Speckle tracking echocardiography — A 24-h ambulatory Holter Echocardiography Speckle tracking echocardiography (STE)

SUMMARY:
Marker of atrial cardiopathay as apredictor value of ischemic stroke

DETAILED DESCRIPTION:
detection of the presence of atrial dysfunction or atrial cardiopathy and its degree among patients complaining of palpitation, with a one-year follow-up for any cardioembolic events (stroke /TIA).

ELIGIBILITY:
Inclusion Criteria:

* Patients complaining of palpitation referred for Holter monitoring

Exclusion Criteria:

* • Valvular AF, moderate to severe mitral/ tricuspid/ aortic stenosis or regurgitation.

  * Recent myocardial infarction within 3 months.
  * Acute pulmonary embolism.
  * Newly onset AF during or shortly after cardiac surgery.
  * Specific type of cardiomyopathy such as cardiac amyloidosis, obstructive hypertrophic cardiomyopathy.

Decompensation stage of organ failure

Ages: 17 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: - Patients complaining of palpitation referred for Holter monitoring
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-11-30 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Detection of any underlying arrythmia after holter monitoring for twenty four hours | Detection of any underlying arrythmia after holter monitoring for twenty four hours
  Detection of any underlying arrythmia after holter monitoring for twenty four hours

SECONDARY OUTCOMES:
Detection of atrial dysfunction or atrial cardiopathy and its degree among patients complaining of palpitation, with 6 month follow-up for any cardioembolic events (stroke /TIA). | Detection of atrial dysfunction or atrial cardiopathy and its degree among patients complaining of palpitation, with 6 month follow-up for any cardioembolic events (stroke /TIA).
  Detection of atrial dysfunction or atrial cardiopathy and its degree among patients complaining of palpitation, with 6 month follow-up for any cardioembolic events (stroke /TIA).

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Aboelkassem Farghal, professor, Principal Investigator — Assiut University
Locations (1):
- Mariam zarief farhan, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided